CLINICAL TRIAL: NCT04850170
Title: The Evaluation of Manual Therapy for the Prevention of Radiation-Induced Fibrosis in Patients With Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202002052A3; CMRPVVL0081 (Other Grant/Funding Number: Chang Gung memorial hospital)
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-04

CONDITIONS: Radiation-Induced Fibrosis in Patients With Head and Neck Cancer
Keywords: Head and neck cancer; Post-radiation fibrosis; Manual therapy; Rehabilitation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Musculoskeletal Manipulations; Speech Therapy

STUDY DESIGN:
Intervention Model Description: The subjects in this study are the patients with head and neck cancer after completion of the radiotherapy. Radiation-induced fibrosis is inevitable and there is no effective treatment to prevent it now. Therefore, there are two parts in this study :
  The first part is a pilot study. There will be 10 subjects included and manual therapy and rehabilitation will be arranged for 6 months. The manual therapy would be once a week at most, and the rehabilitation would be twice a week at most.
  The second part is a randomized controlled study. 60 patients would be randomized divided into two groups. The group 1 is manual therapy(once a week at most) and rehabilitation(twice a week at most), and the group 2 is rehabilitation only(twice a week at most).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The first ten subjects will be enrolled in a pilot study. The following sixty subjects will be separated randomly to experimental group and control group.
  The first ten subjects and the experimental group will be arranged manual therapy and rehabilitation for six months.
  Interventions: Procedure: manual therapy; Procedure: Speech therapy
- Control group (Active Comparator): The control group will be arranged rehabilitation.
  Interventions: Procedure: Speech therapy

INTERVENTIONS:
Procedure: manual therapy — 1. release and stretch the muscles and fascia around shoulder girdle、upper arm and forearm;
  2. massage the masseter muscle and temporalis muscle;
  3. mobilization of the temporomandibular joint, the thoracic and cervical spine, shoulder, and elbow.
  Arms: Experimental group
Procedure: Speech therapy — include the stretching of the neck, facial and oral movement training, and swallowing training

SUMMARY:
The subjects in this study are the patients with head and neck cancer after completion of the radiotherapy. Radiation-induced fibrosis is inevitable and there is no effective treatment to prevent it. Therefore, there are two parts in this study :

The first part is a pilot study. There will be 10 subjects included and manual therapy and rehabilitation will be arranged for 6 months. The manual therapy would be once a week at most, and the rehabilitation would be twice a week at most.

The second part is a randomized controlled study. 60 patients would be randomized divided into two groups. The group 1 is manual therapy(once a week at most) and rehabilitation(twice a week at most), and the group 2 is rehabilitation only(twice a week at most). Patients would be evaluated at baseline, 3rd, 6th, and 12th month. The evaluation is including the degree of superficial soft tissue fibrosis, numerical rating scale of pain, range of motion(neck), range of motion(shoulder), width of mouth opening, EORTC QLQ C30, EORTC QLQ H&N 35, and functional oral intake scale. Besides, swallowing video fluoroscopy would be done at baseline, 6th, and 12th month.

When the subject completes the evaluation in the 12th month, the study is ended.

Because the radiation-induced fibrosis is progressed with time, we will follow up the condition of subjects at the next year and the following third year.

ELIGIBILITY:
Inclusion Criteria :

1. Age > 20 years
2. Head and neck cancer
3. After Completion of radiation therapy for 4 to 6 weeks
4. Be willing to accept manual therapy and long-term follow up

Exclusion Criteria :

1. Recurrence, metastatic cancer, or concurrent second cancer
2. With post-radiation dermatitis at neck or shoulder
3. Current pregnancy or lactation
4. Life expectancy of < 12 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline range of motion, neck at the 3rd month | baseline and 3rd month
  including neck flexion, extension, right and left lateral flexion, and lateral rotation
Change from Baseline Functional oral intake scales at 3rd month | baseline and 3rd month
  in this scales, the maximum values is grade seven, the minimum values is grade one. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
range of motion, shoulder | measure the range of motion at baseline, the 3rd month, the 6th month, the 12th month, the second year, and the third year
  to measure the degree of bilateral shoulder, including flexion, extension, abduction, adduction, external rotation, and internal rotation
Width of mouth opening | at baseline, the 3rd month, the 6th month, the 12th month, the second year, and the third year
  measure the maximum interincisal opening and range of the jaw and mouth
EORTC QLQ C30 | at baseline, the 3rd month, the 6th month, the 12th month, the second year, and the third year
  the most widely used questionnaire for cancer patients; explore aspects of quality of life assessment, evaluation and interpretation.
EORTC H&N 35 | at baseline, the 3rd month, the 6th month, the 12th month, the second year, and the third year
  questionnaire for head and neck cancer patients.
Numerical rating scale of pain | at baseline, the 3rd month, the 6th month, the 12th month, the second year, and the third year
  evaluate the pain degree(0~10); higher scores mean a worse outcome
Swallowing Video Fluoroscopy | at baseline, the 6th month, and the 12th month
  Observe that the patient swallows items with different thicknesses and textures via using a special real-time form of x-ray. This examination allows us to test the ability to swallow safely and effectively.
Change from Baseline range of motion, neck at the the 6th month | baseline and 6th month
  including neck flexion, extension, right and left lateral flexion, and lateral rotation
Change from Baseline range of motion, neck at the the 12th month | baseline and 12th month
  including neck flexion, extension, right and left lateral flexion, and lateral rotation
Change from Baseline range of motion, neck at the the 2nd year | baseline and 2nd year
  including neck flexion, extension, right and left lateral flexion, and lateral rotation
Change from Baseline range of motion, neck at the the 3rd year | baseline and 3rd year
  including neck flexion, extension, right and left lateral flexion, and lateral rotation
Change from Baseline Functional oral intake scales at 6th month | baseline and 6th month
  in this scales, the maximum values is grade seven, the minimum values is grade one. The higher scores mean a better outcome.
Change from Baseline Functional oral intake scales at 12th month | baseline and 12th month
  in this scales, the maximum values is grade seven, the minimum values is grade one. The higher scores mean a better outcome.
Change from Baseline Functional oral intake scales at 2nd year | baseline and 2nd year
  in this scales, the maximum values is grade seven, the minimum values is grade one. The higher scores mean a better outcome.
Change from Baseline Functional oral intake scales at 3rd year | baseline and 3rd year
  in this scales, the maximum values is grade seven, the minimum values is grade one. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- New Taipei Municipal Tucheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang B, Wei J, Meng L, Wang H, Qu C, Chen X, Xin Y, Jiang X. Advances in pathogenic mechanisms and management of radiation-induced fibrosis. Biomed Pharmacother. 2020 Jan;121:109560. doi: 10.1016/j.biopha.2019.109560. Epub 2019 Nov 15. PMID 31739160
- [Background] Purkayastha A, Sharma N, Sarin A, Bhatnagar S, Chakravarty N, Mukundan H, Suhag V, Singh S. Radiation Fibrosis Syndrome: the Evergreen Menace of Radiation Therapy. Asia Pac J Oncol Nurs. 2019 Jul-Sep;6(3):238-245. doi: 10.4103/apjon.apjon_71_18. PMID 31259219
- [Background] Hojan K, Milecki P. Opportunities for rehabilitation of patients with radiation fibrosis syndrome. Rep Pract Oncol Radiother. 2013 Aug 8;19(1):1-6. doi: 10.1016/j.rpor.2013.07.007. eCollection 2014 Jan. PMID 24936313
- [Background] Moloney EC, Brunner M, Alexander AJ, Clark J. Quantifying fibrosis in head and neck cancer treatment: An overview. Head Neck. 2015 Aug;37(8):1225-31. doi: 10.1002/hed.23722. Epub 2014 Jul 11. PMID 24797251
- [Background] Davis AM, Dische S, Gerber L, Saunders M, Leung SF, O'Sullivan B. Measuring postirradiation subcutaneous soft-tissue fibrosis: state-of-the-art and future directions. Semin Radiat Oncol. 2003 Jul;13(3):203-13. doi: 10.1016/S1053-4296(03)00022-5. PMID 12903010
- [Background] Raj VS, Pugh TM, Yaguda SI, Mitchell CH, Mullan SS, Garces NS. The Who, What, Why, When, Where, and How of Team-Based Interdisciplinary Cancer Rehabilitation. Semin Oncol Nurs. 2020 Feb;36(1):150974. doi: 10.1016/j.soncn.2019.150974. Epub 2020 Jan 16. PMID 31955923
- [Background] Krisciunas GP, Vakharia A, Lazarus C, Taborda SG, Martino R, Hutcheson K, McCulloch T, Langmore SE. Application of Manual Therapy for Dysphagia in Head and Neck Cancer Patients: A Preliminary National Survey of Treatment Trends and Adverse Events. Glob Adv Health Med. 2019 Apr 24;8:2164956119844151. doi: 10.1177/2164956119844151. eCollection 2019. PMID 31041144
- [Background] Krisciunas GP, Golan H, Marinko LN, Pearson W, Jalisi S, Langmore SE. A novel manual therapy programme during radiation therapy for head and neck cancer - our clinical experience with five patients. Clin Otolaryngol. 2016 Aug;41(4):425-31. doi: 10.1111/coa.12535. Epub 2016 Feb 8. No abstract available. PMID 26381894